CLINICAL TRIAL: NCT07366788
Title: Evaluation of Dental Pain, Anxiety, and Extraction Efficiency in Mandibular Primary Molar Extraction Using Physics Forceps in Children Aged 6-9 Years: A Randomized Clinical Trial
Brief Title: Clinical Outcomes of Mandibular Primary Molar Extraction Using Physics Forceps in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Principal Investigator, Shadi Azzawi, Head of Pediatric Dentistry Department, Damascus University, Damascus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2324
Record Dates: First submitted 2026-01-09; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Dental Anxiety; Dental Pain; Dental Extraction; Primary Molar Tooth
Keywords: Dental pain; Physics forceps; Conventional forceps; Dental Anxiety; Dental Extraction
MeSH Terms: conditions — Toothache

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This was a double-blind study: both participants and the data analyst were unaware of the group allocations. The children were not informed about their group assignment or the specific aim of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1: Physics forceps - 40 participants. (Active Comparator): - Intervention Arm: Extraction of mandibular primary first and second molars using Physics forceps. Following topical anesthesia with 20% benzocaine gel, local anesthesia was administered using 4% articaine with 1:100,000 epinephrine. Tooth extraction was performed according to the manufacturer's instructions, without conventional rotational movements.
  Interventions: Device: ARM 1 Physics forceps (40 Participant)
- Arm 2: Conventional forceps - 40 participants (Active Comparator): - Control Arm: Extraction of mandibular primary first and second molars using conventional instruments, including periosteal elevators, straight elevators, and conventional pediatric forceps, following standard clinical practice.
  Interventions: Device: ARM 2 conventional forceps (40 Participant)

INTERVENTIONS:
Device: ARM 1 Physics forceps (40 Participant) — After obtaining the child's medical history, clinical and radiographic exams assessed the restorability of lower primary molars and the need for extraction. Written informed consent was obtained from parents/guardians. Participants were randomized using a computer-generated sequence (www.randomization.com). Baseline anxiety was measured via pulse rate and the Facial Image Scale. The procedure was explained using Tell-Show-Do. Topical 20% benzocaine was applied before 4% articaine with 1:100.00 epinephrine. Pain during anesthesia was assessed with FLACC. Post-anesthesia anxiety was reassessed and anesthesia adequacy verified. Tooth extraction was performed with physics ; pain, anxiety, and procedure duration were recorded. Post-extraction, tooth fracture, gingival tearing were evaluated , and postoperative instructions were given
  Arms: Arm 1: Physics forceps - 40 participants.
Device: ARM 2 conventional forceps (40 Participant) — After obtaining the child's medical history, clinical and radiographic exams assessed the restorability of lower primary molars and the need for extraction. Written informed consent was obtained from parents/guardians. Participants were randomized using a computer-generated sequence (www.randomization.com). Baseline anxiety was measured via pulse rate and the Facial Image Scale. The procedure was explained using Tell-Show-Do. Topical 20% benzocaine was applied before 4% articaine with 1:100.00 epinephrine. Pain during anesthesia was assessed with FLACC. Post-anesthesia anxiety was reassessed and anesthesia adequacy verified. Tooth extraction was performed by conventional forceps; pain, anxiety, and procedure duration were recorded. Post-extraction, tooth fracture, gingival tearing were evaluated , and postoperative instructions were given
  Arms: Arm 2: Conventional forceps - 40 participants

SUMMARY:
Tooth extraction is a common procedure and often associated with pain, fear, and discomfort especially in pediatric patients, which may lead to a negative attitude toward the dental. Therefore, identifying techniques that reduce pain and anxiety while improving procedural efficiency is of clinical importance.

This randomized clinical trial aimed to evaluate the efficiency of Physics forceps on dental pain, anxiety, and extraction in children aged 6-9 years undergoing primary molar extraction.

Eligible children requiring extraction of lower primary molars will be randomly assigned to one of two groups based on the type of extraction forceps used (Physics or conventional).

Dental anxiety will be assessed using both physiological measures (pulse rate) and subjective measures (Facial Image Scale).

Pain perception will be evaluated using the FLACC pain scale during local anesthesia administration and tooth extraction.

The duration of the extraction procedure will be recorded, and any intraoperative complications will be documented.

The findings of this study provide clinical evidence regarding the effectiveness of Physics forceps in reducing pain and anxiety and improving extraction efficiency among pediatric patients in a dental clinic, which leads to better clinical decision-making and enhanced pediatric patient care.

DETAILED DESCRIPTION:
This study investigates the use of a physics forceps compared with a conventional forceps during the extraction of mandibular primary molars in pediatric dental patients. Extraction of primary molars is a frequently performed procedure in pediatric dentistry and is often associated with dental anxiety, pain perception, and behavioral management challenges. Improving extraction techniques may positively influence the child's experience as well as the clinician's efficiency.

The study focuses on evaluating whether the use of a physics forceps can contribute to a more favorable clinical and patient-centered outcome when compared to traditional extraction instruments. The intervention does not introduce any additional or experimental dental procedures, as all tooth extractions included in the study are clinically indicated and performed as part of routine dental care.

The comparison between the two extraction approaches aims to assess their impact on child comfort, emotional response during treatment, and procedural efficiency. Particular attention is given to outcomes related to pain perception, anxiety levels, and the overall duration of the extraction procedure, as these factors play a significant role in pediatric dental management.

In addition to patient-centered outcomes, the study also considers operator-related and procedural aspects, including ease of use and the occurrence of intraoperative difficulties or complications. All clinical procedures are carried out following standard pediatric dental protocols, ensuring that patient safety and ethical principles are fully respected.

Data collected from this study are intended to provide clinically meaningful insight into whether Physics forceps offer advantages over conventional forceps in routine pediatric dental practice. The results may support evidence-based decision-making when selecting extraction instruments for children and may contribute to improving the overall quality of care during primary tooth extraction.

ELIGIBILITY:
Inclusion Criteria:

For both groups, the inclusion criteria were:

1. Children aged 6 - 9 years.
2. Healthy children with no history of neurological disorders or systemic diseases.
3. Mandibular primary molars indicated for extraction, with at least half of the root length remaining.
4. Cooperative behavior classified as Frankl 3 - 4.
5. Absence of acute inflammation or active periapical/periodontal infection at the time of extraction

Exclusion Criteria:

- 1. Children who were taking medications that may alter pain perception or bleeding tendency.

2. Teeth with insufficient root structure that made extraction technically unfeasible.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2025-05-21 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Dental pain | During local anesthesia administration (from needle insertion until needle withdrawal). During tooth extraction (from forceps application on tooth until tooth removal).
  Pain intensity assessed using FLACC behavioral observational scale (Face, Legs, Activity, Cry, Consolability), with a total score from 0 to 10(0 = Relaxation, 1 - 3 = Mild discomfort, 4 - 6 = Moderate discomfort, 7 - 10 = Severe discomfort
Extraction Time | Periprocedurally (during extraction),from the second the forceps is applied on the tooth until the second the tooth is out.
  Duration of extraction procedure measured from forceps application until complete removal of the tooth. - Unit of Measure: Seconds.

SECONDARY OUTCOMES:
Dental Anxiety - Pulse Rate | - Baseline (upon seating, before procedure). - After local anesthesia administration. - During extraction.
  Anxiety assessed objectively by pulse rate using pulse oximeter. Unit of Measure: Beats per minute (bpm)
Dental Anxiety - Facial Image Scale (FIS) | - Baseline (upon seating, before procedure). - After local anesthesia administration. - Immediately after extraction.
  Anxiety assessed subjectively using Facial Image Scale (score 1-5), very happy (score =1) to very unhappy (score =5).
Intraoperative Complications | Immediately after extraction.
  Presence or absence of tooth fracture and/or soft tissue tearing documented on structured data collection form.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatric Dentistry - Prof. Shadi Azzawi., Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Laskar S, Singh M, Suman A, Sahu S, Mishra BP, Sahoo A. Efficacy of the Atraumatic Physics Forceps Over Conventional Extraction Forceps in Extraction of Tooth-Does it Offer an Alternative in All Types of Extraction or Only can be Used in Few Selected Types of Extraction: A Comparative Study. J Pharm Bioallied Sci. 2022 Jul;14(Suppl 1):S859-S862. doi: 10.4103/jpbs.jpbs_27_22. Epub 2022 Jul 13. PMID 36110718
- [Result] Mutashar HA, Abdulrazaq SS. Evaluation and Comparison of Physics Forceps and Conventional Forceps in Bilateral Dental Extraction: A Randomized, Split-Mouth, Clinical Study. Cureus. 2023 Apr 27;15(4):e38206. doi: 10.7759/cureus.38206. eCollection 2023 Apr. PMID 37252611
- [Result] Kapila S, Kaur T, Bhullar RS, Sandhu A, Dhawan A, Kaur A. Use of Physics Forceps in Atraumatic Orthodontic Extractions of Bilateral Premolars: A Randomized Control Clinical Study. J Maxillofac Oral Surg. 2020 Sep;19(3):347-354. doi: 10.1007/s12663-020-01347-6. Epub 2020 May 5. PMID 32801526
- [Result] Hariharan S, Narayanan V, Soh CL. Split-mouth comparison of physics forceps and extraction forceps in orthodontic extraction of upper premolars. Br J Oral Maxillofac Surg. 2014 Dec;52(10):e137-40. doi: 10.1016/j.bjoms.2014.06.013. Epub 2014 Jul 8. PMID 25015020
- [Result] Elicherla SR, Bandi S, Nunna M, Saikiran KV, Sahithi V, Nuvvula S. Comparative evaluation of efficacy of Physics Forceps versus conventional forceps in pediatric dental extractions: a prospective randomized study. J Dent Anesth Pain Med. 2021 Dec;21(6):547-556. doi: 10.17245/jdapm.2021.21.6.547. Epub 2021 Nov 26. PMID 34909472